CLINICAL TRIAL: NCT05161715
Title: A Phase 2a, Proof-of-Concept, Open-Label Study to Evaluate the Pharmacodynamics, Pharmacokinetics, and Safety of Obicetrapib in Patients With Early Alzheimer's Disease (Hetero/Homozygote APOE4 Carriers)
Brief Title: Proof-of-concept, Open-label Study in Patients With Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TA-8995 AD-1
Record Dates: First submitted 2021-11-23; First posted 2021-12-17 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-10

CONDITIONS: Early Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — TA-8995

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 10mg obicetrapib tablets (Experimental): 10mg obicetrapib (5mg tablets) administered orally daily for 24 weeks
  Interventions: Drug: Obicetrapib

INTERVENTIONS:
Drug: Obicetrapib — 10mg obicetrapib
  Other Names: TA-8995

SUMMARY:
A Phase 2a study in men and women with early Alzheimer's disease to evaluate the pharmacodynamics, pharmacokinetics and safety of obicetrapib therapy.

DETAILED DESCRIPTION:
This study will be a proof of concept, Phase 2a study in patients with early Alzheimer's disease (clinical diagnosis of Alzheimer's disease Stage 3 or 4 based on the National Institute on Aging Alzheimer's Association Research Framework criteria) to evaluate the Pharmacodynamic, cognitive effects, Pharmacokinetic, and safety and tolerability of obicetrapib therapy.

ELIGIBILITY:
Inclusion Criteria:

* men & women 50-75 years
* post-menopausal or women not of child-bearing potential
* diagnosis of Alzheimer's disease based on National Institute for Aging:
* Biomarker classification A+T+N+ or A+T+N-
* Clinical Stage 3 or 4 with Clinical Dementia Rating score >/= 0.5 & </= 1; mini-mental state examination (MMSE) score >/=20
* Have an APOE genotype of E4/E4 or E3/E4
* not on or on stabilized AD medication
* Patient & study partner willing to sign consent

Exclusion Criteria:

* Other than AD, disorder that may impair cognition
* Contra-indication for MRI
* History of neurological, psychiatric or mental conditions;

  * history stroke
  * MI
  * Type 1 diabetes & Type 2 with HbA1c>8%
  * BP > 150/90 mmHg
  * renal or hepatic impaired
  * hyperaldosteronism
  * cancer
  * depression
  * laboratory abnormalities
  * not able to undergo lumbar puncture
  * taking certain medications including lipid altering

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ditmarsch, MD, Study Director — NewAmsterdam Pharma
Locations (1):
- Brain Research Center Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 10mg Obicetrapib: 10mg obicetrapib (5mg tablets) administered orally daily for 24 weeks
  Obicetrapib: 10mg obicetrapib
Period: Overall Study
Arm/Group | 10mg Obicetrapib
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline Population is defined as all participants who received at least one dose of study drug.
Arm/Group | 10mg Obicetrapib
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Apolipoprotein A-I (ApoA-I) in Cerebrospinal Fluid (CSF)
Description: Mean percent change from screening (V1) to end of treatment (V6) in ApoA-I in CSF
Time Frame: 24 weeks
Population: Analysis of PD endpoints in CSF were conducted on 12 patients as the lumbar puncture for one patient was unsuccessful at End of Treatment (Day 168, Visit 6) and no CSF was available for analysis.
Measure: Mean (Standard Deviation); unit: percent change from screening visit
Arm/Group | 10mg Obicetrapib
Number analyzed (Participants) | 12
percent change from screening visit | -8.4 (13.6)
Statistical Analysis 1: Comparison: 10mg Obicetrapib; Test type: Other; p = 0.425, Wilcoxon (Mann-Whitney) — No multiple testing correction was performed

2. Primary Outcome: Mean Percent Change in Apolipoprotein A-I (ApoA-I) in Plasma
Description: Mean percent change in ApoA-I in plasma from baseline (V2) to week 24 (V6)
Time Frame: 24 weeks
Population: For the PD endpoints in plasma, analyses were conducted on all 13 patients.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | 10mg Obicetrapib Tablets
Number analyzed (Participants) | 13
percent change from baseline | 37.5 (25.2)
Statistical Analysis 1: Comparison: 10mg Obicetrapib Tablets; Test type: Other; p = 0.0002, Wilcoxon (Mann-Whitney) — No multiple testing correction was performed

3. Primary Outcome: Mean Percent Change in Apolipoprotein-E (ApoE) in Cerebrospinal Fluid (CSF)
Description: Mean percent change from screening (V1) to end of treatment (V6) in ApoE
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from screening
Arm/Group | 10mg Obicetrapib Tablets
Number analyzed (Participants) | 12
percent change from screening | 3.9 (10.3)
Statistical Analysis 1: Comparison: 10mg Obicetrapib Tablets; Test type: Other; p = 0.0424, Wilcoxon (Mann-Whitney) — No multiple testing correction was performed

4. Primary Outcome: Mean Percent Change in Apolipoprotein-E (ApoE) in Plasma
Description: Mean percent change from baseline (V2) to week 24 (V6) in plasma in ApoE
Time Frame: 24 weeks
Population: For the PD endpoints in plasma, analyses were conducted on all 13 patients.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | 10mg Obicetrapib Tablets
Number analyzed (Participants) | 13
percent change from baseline | 47.8 (46.9)
Statistical Analysis 1: Comparison: 10mg Obicetrapib Tablets; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney) — No multiple testing correction was performed

5. Primary Outcome: Small HDL (s-HDL) Particle Concentration in Cerebrospinal Fluid (CSF) at Baseline
Description: Small high-density lipoprotein (s-HDL) particle concentration in cerebrospinal fluid (CSF) measured by Ion Mobility Assay (https://doi.org/10.1002/alz.12649)
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average relative abundance
Arm/Group | 10mg Obicetrapib Tablets
Number analyzed (Participants) | 12
average relative abundance | 0.542 (0.138)

6. Primary Outcome: Small HDL (s-HDL) Particle Concentration in Cerebrospinal Fluid (CSF) at Week 24
Description: Small high-density lipoprotein (s-HDL) particle concentration in CSF measured by Ion Mobility Assay (https://doi.org/10.1002/alz.12649)
Time Frame: Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average relative abundance
Arm/Group | 10mg Obicetrapib Tablets
Number analyzed (Participants) | 12
average relative abundance | 0.542 (0.106)

7. Primary Outcome: Small HDL (s-HDL) Particle Concentration in Plasma at Baseline
Description: Small high-density lipoprotein (s-HDL) particle concentration plasma measured by Ion Mobility Assay.
  For more information on the measurement used please refer to this article: https://doi.org/10.1002/alz.12649
Time Frame: baseline
Population: Due to a non-optimal sample preparation procedure, a number of the samples allocated for the small HDL-C particle analysis were lost and therefore no samples were assessed for this measure.
Arm/Group | 10mg Obicetrapib
Number analyzed (Participants) | 0

8. Primary Outcome: Small HDL (s-HDL) Particle Concentration in Plasma at Week 24
Description: Small high-density lipoprotein (s-HDL) particle concentration in plasma measured by Ion Mobility Assay at Week 24
  For more information on the measurement used please refer to this article: https://doi.org/10.1002/alz.12649
Time Frame: Week 24
Population: as for outcome 7
Arm/Group | 10mg Obicetrapib
Number analyzed (Participants) | 0

9. Primary Outcome: Mean Percent Change in Cholesterol Efflux Capacity in Cerebrospinal Fluid (CSF)
Description: Mean percent change in cholesterol efflux capacity in CSF from screening (V1) to week 24 (V6)
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from screening
Arm/Group | 10mg Obicetrapib Tablets
Number analyzed (Participants) | 12
percent change from screening | 1.9 (24.1)
Statistical Analysis 1: Comparison: 10mg Obicetrapib Tablets; Test type: Other; p = 0.556, Wilcoxon (Mann-Whitney) — No multiple testing correction was performed

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Week 24.5
Description: Safety Population included all participants who received at least 1 dose of any study drug.
  Analysis of PD endpoints in CSF were conducted on 12 patients as the lumbar puncture for one patient was unsuccessful at End of Treatment (Day 168, Visit 6) and no CSF was available for analysis. For the PD endpoints in plasma, analyses were conducted on all 13 patients.
Arm/Group | 10mg Obicetrapib Tablets
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10mg Obicetrapib Tablets (N=13)
Normocytic anemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Benign paroxysmal positional vertigo (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Loose stools (Gastrointestinal disorders) | 1 (1)
Obstipation (Gastrointestinal disorders) | 1 (1)
Reflux esophagitis (Gastrointestinal disorders) | 1 (1)
Unilateral leg swelling (General disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Lumbar puncture headache (Injury, poisoning and procedural complications) | 1 (1)
Rib contusion (Injury, poisoning and procedural complications) | 1 (1)
Weight loss (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hand arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lateral epicondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbago (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma face (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 12 months after completion of the study, whichever occurs first, Institution may publish the results of its study data. Institution and PI shall provide Sponsor with an advance copy of any proposed communications at least 30 days prior and Sponsor shall have 30 days to review. Sponsor may request (a) the deletion of any Confidential Information, (b) reasonable changes, or (c) a delay for an additional 60 day period.

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT05161715/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT05161715/SAP_001.pdf